CLINICAL TRIAL: NCT04857567
Title: The Efficacy Study of the Evidence-Based Psychological Intervention for Improving Resilience and Preventing Burnout of Residents
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: Mind Works Clinical Psychologist Group (Unknown)
Responsible Party: Principal Investigator, Heung-Kwon Oh, Clinical Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: B-2007/624-304
Record Dates: First submitted 2021-04-07; First posted 2021-04-23 (Actual); Last update posted 2021-07-28 (Actual); Status verified 2021-07

CONDITIONS: Burn Out (Psychology)
Keywords: resident; surgery; ego resilience; mindfulness
MeSH Terms: conditions — Burnout, Psychological

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Three Self-Commitment (TSC) program (Experimental)
  Interventions: Behavioral: TSC program (Three Self-Commitment program)

INTERVENTIONS:
Behavioral: TSC program (Three Self-Commitment program) — 1. Self-Competence program
     - A program for residents who experience exhaustion due to the spirit of volunteerism and high expectations of therapeutic competency in the case of experiencing a decrease in personal achievement.
  2. Self-Care program
     - A program to help individuals who experience dehumanization due to emotional suppression and develop exhaustion in the process of suppressing emotions to protect themselves from excessive feelings of compassion experienced in the medical scene
  3. Self-Compassion program - A program for residents who experience emotional burnout and exhaustion due to pressure of failure because medical professionals should be competent and excellent

SUMMARY:
There are few systematic studies on the working environment and mental health of residents who are at the forefront of Korean medical care. In particular, there is no scientific research on burnout prevention. Since preventing burnout of surgical residents is directly related not only to personal well-being but the health of the patients, it is necessary to care for the individual's psychological state at a social level. This psychological intervention program that is expected to improve recovery resilience in stressful situations of residents and prevent burnout is implemented, and its effectiveness is to be verified.

ELIGIBILITY:
Inclusion Criteria:

* Surgical trainees (residents and clinical fellows) at Bundang Seoul National University Hospital, who is 20 years of age or older, regardless of sex or race.

Exclusion Criteria:

* Subjects who do not consent to the study
* Subjects with meditation experience

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
TCI, Temperament and Character Inventory | Change from baseline at right after 6 cycles of TSC program (up to 24 weeks from baseline)
  A test developed by Clononger, Przybeck, Svrakic and Wetzel (1994) and currently widely used in various countries such as the United States, France, and Spain.
  A tool that measures personality traits such as autonomy, solidarity, and self-transcendence, along with individual traits such as stimulation seeking, risk aversion, social sensitivity, and endurance. In this study, the Korean version (Min et al., 2007) of the German version of TCI-RS, the standardized test, is adapted : Based on the test result, the individual's personality characteristics of the resident are identified and applied.
MBI, Maslach Burnout Inventory | Change from baseline at right after 6 cycles of TSC program (up to 24 weeks from baseline)
  As a test developed by Maslach and Jackson (1981), MBI is a tool that measures the sub-concepts of burnout, such as emotional burnout, dehumanization, and personal sense of accomplishment.
  MBI is a measurement tool used in more than 90% of empirical exhaustion research worldwide, and a test developed to measure the exhaustion of personnel providing interpersonal services including medical workers.
  In this study, MBI adapted and validated by Kang Jeong-hee and Kim Cheol-woong (2012) is used. Participate in the program according to the type of burnout of the client and measure the change in the burnout level of the participants before and after.
ER89, Ego Resilience Scale | Change from baseline at right after 6 cycles of TSC program (up to 24 weeks from baseline)
  A test developed by Block and Kremen (1996) that measures sub-concepts of self-elasticity such as interpersonal relationships, vitality, emotional control, curiosity, and optimism.
  In this study, a scale adapted by Park Eun-hee (1997), which was verified as 76-79, is used and measures the change in the participant's ego-elasticity before and after participating in the program.
DASS-21, Depression Anxiety StressScale | In this study, changes in participant's psychological pain are measured at each session during the program (6 cycles of TSC program, 3-4 weeks interval, up to 24 weeks from baseline).
  A test developed by Lovibond and Lovibond (1995) to measure depression, anxiety, and stress corresponding to psychological distress.
  The internal agreement was verified as 0.87~0.91, 0.83~0.89, and 0.83~0.92 for depression, anxiety, and stress, respectively (Youngsun Lee et al, 2019; Jun et al, 2018).
Subjective Well-being | Change from baseline at right after 6 cycles of TSC program (up to 24 weeks from baseline)
  A test developed by Diener E (1985) to measure subjective satisfaction with daily life.
  A tool showing the internal consistency reliability of 0.87 and the test-retest reliability of 0.82.
SCS, Self-Compassion Scale | Change from baseline at right after 6 cycles of TSC program at the end of Cycle 6 (each cycle is 4 weeks, up to 24 weeks from baseline)
  Developed by Neff (2003) and validated as a Korean version by Kim et al. (2008) / 26 items / 6 sub-factors: self-kindness, self-judgment, universal humanity, isolation, mindfulness, hyper-identification on a 5-point scale (minimum 6 to maximum 30, the higher the score, the better the outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Heung-Kwon Oh, PhD, Principal Investigator — Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: Undecided